CLINICAL TRIAL: NCT05486884
Title: Mean Arterial Pressure After Out-of-hospital Cardiac Arrest: the METAPHORE Randomized Trial
Brief Title: Mean Arterial Pressure After Out-of-hospital Cardiac Arrest
Acronym: METAPHORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHM-2022/S03/07
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest; Out-of-hospital Cardiac Arrest (OHCA)
Keywords: cardiac arrest; outcome; cerebral blood flow; mean arterial pressure
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled, open study
Who Masked: Outcomes Assessor
Masking Description: Score mRS will be measured by a psychologist during a telephone interview 180 days after inclusion. The psychologist will be blinded to the randomization arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high MAP threshold (Experimental): Norepinephrine will be titrated to maintain MAP ≥ 90 mmHg. This threshold will be maintained for the 24 hours following inclusion by the perfusion of norepinephrine at an appropriate dose.
  From 24 hours after inclusion until ICU discharge, a MAP ≥ 65 mmHg will be targeted
  Interventions: Procedure: Maintain MAP ≥ 90 mmHg
- standard MAP threshold (Active Comparator): Norepinephrine will be titrated to maintain MAP ≥ 65 mmHg. This target MAP will be maintained for 24 hours after randomization through the perfusion of norepinephrine at an appropriate flow rate.
  From 24 hours after inclusion until ICU discharge, a MAP ≥ 65 mmHg will be targeted
  Interventions: Procedure: Maintain MAP ≥ 65 mmHg

INTERVENTIONS:
Procedure: Maintain MAP ≥ 90 mmHg — Maintain MAP ≥ 90 mmHg for the 24 hours following inclusion by perfusion of norepinephrine
  Arms: high MAP threshold
Procedure: Maintain MAP ≥ 65 mmHg — Maintain MAP ≥ 65 mmHg for 24 hours after randomization through the perfusion of norepinephrine
  Arms: standard MAP threshold

SUMMARY:
Out-of-hospital cardiac arrest is a public health problem for which overall survival is below 10%. Post-cardiac arrest syndrome is the principal cause of death in intensive care units (ICU), due to refractory shock or brain injuries secondary to anoxia. Brain anoxia is responsible for severe neurological sequelae that may be aggravated by cerebral hypoperfusion during the first few hours after the return of spontaneous circulation. Current recommendations are to ensure that arterial blood pressure is sufficient for the perfusion of organs, but no minimum threshold mean arterial pressure (MAP) has been defined. In practice, most teams target a MAP of at least 65 mmHg. Several observational studies have shown a correlation between MAP and neurological prognosis, patients with a higher initial MAP having a better outcome. Recent pilot studies have demonstrated the feasibility of increasing the target MAP after cardiac arrest, but conflicting results have been obtained concerning patient prognosis. These findings may be explained by changes to the autoregulation of the brain after cardiac arrest, with a shift of the curve towards the right, or its abolition. Cerebral blood flow is dependent on MAP, and a target MAP of 65 mmHg for these patients may result in insufficient brain perfusion. Conversely, a too high MAP might cause brain lesions due to vasogenic edema, hemorrhagic complications or excess perfusion in conditions of diminished brain metabolism. An interventional study is required to evaluate the effect of increasing MAP on neurofunctional outcome after cardiac arrest. Given the data available for brain autoregulation, the correlation between MAP and prognosis, and the risks theoretically associated with a higher MAP, investigator plans to compare a standard threshold of MAP (≥ 65 mmHg) with a high threshold of MAP (≥ 90 mmHg). Investigator hypothesizes that a high MAP within the first 24 hours after cardiac arrest will improve neurofunctional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU following an out-of-hospital cardiac arrest with an initially shockable or non-shockable rhythm ;
* Sustained ROSC defined as 20 minutes with signs of circulation without the need for chest compressions;
* Under invasive mechanical ventilation for coma, defined as a Glasgow score ≤ 8/15;
* Consent from a relative or of a procedure for emergency inclusion.

Exclusion Criteria:

* Age < 18 years ;
* In-hospital cardiac arrest (first cardiac arrest);
* Unwitnessed CA with initial rhythm of asystole
* Delay between ROSC and attempting randomisation > 6 hours ;
* Cardiac arrest in a context of multiple trauma ;
* Cardiac arrest in a context of hemorrhagic shock or severe hemorrhage necessitating hemostasis (surgery or radiological or endoscopic hemostasis) ;
* Cardiac arrest secondary to an acute brain disease (ischemic or hemorrhagic stroke, subarachnoid hemorrhage, severe traumatic brain injury) ;
* Refractory shock :

Defined as a MAP < 65 mmHg for more than one hour on norepinephrine or epinephrine at a dose > 1 µg/kg/min despite adequate fluid resuscitation ;

* Extracorporeal circulatory support prior to inclusion;
* Known allergy to norepinephrine or to any of its excipients;
* Decision to limit care before inclusion ;
* Modified Rankin score of 4 or 5 before cardiac arrest ;
* Inclusion in another interventional study in which the principal endpoint is neurological prognosis ;
* Pregnancy or breast feeding ;
* Adult patient deprived of freedom or under legal protection (patients under guardianship or curatorship) (article L1121-6 of the French Health Code) ;
* Non-French speaking;
* Patient already included in this trial ;
* Absence of social security cover.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a good neurofunctional outcome 180 days after inclusion | 180 days after inclusion
  Good neurofunctional outcome will be defined by a modified Rankin scale (mRS) of 0 to 3.This score is a global evaluation scale for disability, with seven levels (0 = no symptoms; 6 = patient dead).This score will be measured by psychologist who will be blinded to the randomization arm.

SECONDARY OUTCOMES:
Proportion of patients alive at Intensive Care Unit discharge, at hospital discharge, at day 28 (D28) and six months (D180) after inclusion | From Intensive Care Unit admission to Intensive Care Unit discharge (up to 3 weeks), from hospital admission to hospital discharge (up to 12 weeks), 28 days and 180 days after inclusion
  Proportion of patients alive at Intensive Care Unit discharge, at hospital discharge, at day 28 (D28) and six months (D180) after inclusion
Proportion of patients alive at Intensive Care Unit discharge with good neurofunctionnal outcome | From Intensive Care Unit admission to Intensive Care Unit discharge (up to 3 weeks)
  Good neurofunctional outcome will be defined by a modified Rankin scale (mRS) of 0 to 3.This score is a global evaluation scale for disability, with seven levels (0 = no symptoms; 6 = patient dead
Quality of life six months after inclusion | 6 months after inclusion
  Quality of life is measured by EuroQol-5D-5L. It's a measure of health-related quality of life and comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). EuroQol-5D-5L could be administered by telephone
Evaluation of Clinical Frailty at six months after inclusion | Six months after inclusion
  Clinical Frailty is measured by the Clinical Frailty Scale (CFS). It summarizes the overall level of fitness or frailty of a patient with a score from 1 (very fit) to 9 (terminally ill)
Number of ICU-free days at Day 28 | Day 28
  Number of ICU-free days is calculated from the number of days alive outside the ICU by Day 28
Number of ventilator-free days, number of catecholamine-free days and number of renal replacement therapy-free days at day 28 | 28 days after inclusion
  Number of ventilator-free days, number of catecholamine-free days and number of renal replacement therapy-free days is calculated from the number of days alive without invasive mechanical ventilation, catecholamine infusion or renal replacement therapy by Day 28
Proportion of patients with acute kidney injury stage 3 and need for renal replacement therapy (RRT) within Intensive Care Unit stay and persistant need for RRT at Intensive Care Unit discharge | From Intensive Care Unit admission to Intensive Care Unit discharge (up to 3 weeks)
  Acute kidney injury stage 3 is defined by at least one of the following criteria: serum creatinine concentration of more than 4 mg/dl (354 µmol/liter) or greater than 3 times the baseline creatinine level, anuria (urine output of 100 ml/day or less) for more than 12 hours, oliguria (urine output below 0.3 ml/kg/h or below 500 ml/day) for more than 24 hours;

OTHER OUTCOMES:
Cardiovascular complications | within 7 days after inclusion
  Cardiovascular complications are assessed by determining the number of patients presenting a severe cardiovascular complication within 7 days of inclusion
Neurological complications | within 7 days of inclusion
  Neurological complications are asssessed by determining the number of patients presenting stroke (ischemic stroke, subarachnoid hemorrhage or cerebral hematoma), confirmed by imaging (CT-scan or MRI) within 7 days of inclusion (systematic cerebral imaging is not required by the protocol but only in case of clinical suspicion of stroke or for neuroprognostication)
Cutaneous complications within 7 days of inclusion | within 7 days of inclusion
  Cutaneous complications are assessed by determining the number of patients presenting necrosis of the extremities within 7 days of inclusion
Digestive complications within 7 days after inclusion | within 7 days of inclusion
  Digestive complications are assessed by determining the number of patients presenting a clinical suspicion of digestive ischemia, confirmed by imaging (CT-scan), endoscopy or exploratory laparotomy, within 7 days of inclusion
Major bleeding within 7 days of inclusion | within 7 days of inclusion
  Major bleeding is assessed by determining the number of patients presenting one of the International Society on Thrombosis and Haemostasis (ISTH) criteria within 7 days of inclusion (fatal bleeding and/or symptomatic bleeding in a critical area or in an organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular, pericardial or intramuscular with compartment syndrome and/or bleeding causing a fall in hemoglobin level of 20 g.L-1 or more or leading to transfusion of two or more units of red cells)
Global complications within 7 days of inclusion | within 7 days of inclusion
  Global complications are defined by the proportion of patients with at least one complication (cardiovascular, neurological, cutaneous, digestive or hemorrhagic) within 7 days of inclusion
Proportion of patients with a good neurofunctional prognosis at six months in the subgroup of patients with an initial shockable cardiac arrest rhythm and in the subgroup of patients with an initial non-shockable cardiac arrest rhythm | 6 months after inclusion
  Proportion of patients with a good neurofunctional prognosis at six months in the subgroup of patients with an initial shockable cardiac arrest rhythm and in the subgroup of patients with an initial non-shockable cardiac arrest rhythm
Proportion of patients with a good neurofunctional prognosis at six months in the subgroup of patients with confirmed chronic arterial hypertension and in the subgroup of patients without chronic arterial hypertension | 6 months after inclusion
  Proportion of patients with a good neurofunctional prognosis at six months in the subgroup of patients with confirmed chronic arterial hypertension and in the subgroup of patients without chronic arterial hypertension. Chronic high blood pressure is defined as need for chronic treatment prior to cardiac arrest;
Proportion of patients with good neurofunctional prognosis at six months in the three risks subgroups of patients identified by CAHP score (< 150, 150-200 and > 200). | 6 months after inclusion
  Proportion of patients with good neurofunctional prognosis at six months in the three risks subgroups of patients identified by CAHP score (< 150, 150-200 and > 200). The CAHP score represents a simple tool for early stratification of patients admitted in ICU after OHCA, using seven variables (age, rhythm, time from collapse to basic life support, time from basic life support to ROSC, location of cardiac arrest, epinephrine dose and arterial pH)

CONTACTS AND LOCATIONS:
Locations (27):
- France (27):
  - CHU Brest - Hôpital de La Cavale Blanche, Brest
  - CH Brive, Brive-la-Gaillarde
  - CHU Caen, Caen
  - CH Cholet, Cholet
  - CH Dieppe, Dieppe
  - CHU Dijon - Hôpital F. Mitterrand, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - CH Versailles, Le Chesnay
  - Centre Hospitalier Du Mans, Le Mans
  - CH Dr Schaffner, Lens
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - APHM - Hôpital de la Timone, Marseille
  - Hôpital Jacques Cartier, Massy
  - CHU Nantes, Nantes
  - CHU Nice - Hôpital Pasteur, Nice
  - CHU Nice - Hôpital Archet, Nice
  - CHU Nîmes, Nîmes
  - CHR Orléans, Orléans
  - Hôpital Cochin, Paris
  - APHP - Hôpital Européen Georges Pompidou (HEGP), Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - Centre Cardiologique du Nord, Saint-Denis
  - CHRU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHRU Tours - Hôpital Bretonneau, Tours
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Yes
After publication of the main results, the anonymized data necessary for carrying out additional analyses may be made available upon request addressed to the coordinating investigator and the scientific committee

REFERENCES:
- [Derived] Chudeau N, Saulnier P, Parot-Schinkel E, Lascarrou JB, Colin G, Barbar SD, Painvin B, Pichon N, Du Cheyron D, Marchalot A, Jarousseau F, Delbove A, Morichau-Beauchant T, Girardie P, Salmon Gandonniere C, Thille AW, Quenot JP, Bailly P, Goudelin M, Martino F, Nigeon O, Merdji H, Brechot N, Bourenne J, Bougouin W, Muller G, Jozwiak M, Doyen D, Rouanet E, Cariou A, Guitton C; AfterROSC Network; CRICS TRIGGERSep F-CRIN Network. Mean arterial pressure after out-of-hospital cardiac arrest (METAPHORE): study protocol for a multicentre controlled trial with blinded primary outcome assessor. BMJ Open. 2025 Apr 25;15(4):e096997. doi: 10.1136/bmjopen-2024-096997. PMID 40280607